CLINICAL TRIAL: NCT06930664
Title: A Phase 1 Clinical Study in Healthy Females of Nonchildbearing Potential to Compare the Pharmacokinetics of Sotatercept (MK-7962) Administered as a Liquid Formulation in an Autoinjector Versus the Lyophilized Formulation
Brief Title: A Study of Sotatercept (MK-7962) in Healthy Females Administered as a Liquid Formulation in an Autoinjector Versus the Lyophilized Formulation (MK-7962-027)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 7962-027; MK-7962-027 (Other: MSD)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose Subcutaneous Injection (Active Comparator): Participants will receive a single subcutaneous high dose of sotatercept administered via syringe.
  Interventions: Biological: Sotatercept
- High Dose Subcutaneous Autoinjector (Experimental): Participants will receive a single subcutaneous high dose of sotatercept administered via autoinjector.
  Interventions: Biological: Sotatercept Autoinjector
- Low Dose Subcutaneous Autoinjector (Experimental): Participants will receive a single subcutaneous low dose of sotatercept administered via autoinjector.
  Interventions: Biological: Sotatercept Autoinjector

INTERVENTIONS:
Biological: Sotatercept — Subcutaneous Injection
  Other Names: MK-7962; ActRIIA-IgG1Fc; ACE-011
  Arms: High Dose Subcutaneous Injection
Biological: Sotatercept Autoinjector — Subcutaneous Auto Injection
  Other Names: MK-7962; ActRIIA-IgGIFc; ACE-011
  Arms: High Dose Subcutaneous Autoinjector; Low Dose Subcutaneous Autoinjector

SUMMARY:
The goal of the study is to learn what happens to different forms of sotatercept medications in a healthy person's body over time. Researchers want to know if there is a difference in the healthy person's body when different forms of sotatercept medications are given.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body weight between 75 and 100 kg, inclusive
* Is assigned female sex at birth and is a participant of nonchildbearing potential (PONCBP) defined as one of the following:

  * Premenarchal
  * Premenopausal with documented hysterectomy and/or bilateral salpingectomy
  * Postmenopausal
  * Medical cause of permanent infertility (eg, Müllerian agenesis, androgen insensitivity)

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of opportunistic infection (eg, invasive candidiasis or pneumocystis pneumonia)
* Has had a serious local infection (eg, cellulitis, abscess) or systemic infection (eg, septicemia) within 3 months prior to screening

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of Sotatercept at High Dose | Predose and at designated timepoints (up to approximately 120 days postdose)
  Blood samples will be collected to determine the AUC0-inf of sotatercept in plasma.
Area Under the Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Sotatercept at High Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the AUC0-last of sotatercept in plasma.
Maximum Observed Concentration (Cmax) of Sotatercept at High Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the Cmax of sotatercept in plasma.

SECONDARY OUTCOMES:
Time of the Maximum Observed Concentration (Tmax) of Sotatercept High Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the Tmax of sotatercept in plasma.
Apparent Terminal Elimination Half-Life (t1/2) of Sotatercept at High Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the t1/2 of sotatercept in plasma.
Apparent Total Plasma Clearance (CL/F) of Sotatercept at High Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the CL/F of sotatercept in plasma.
Apparent Volume of Distribution During Terminal Elimination Phase (Vz/F) of Sotatercept at High Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the Vz/F of sotatercept in plasma.
Cmax of Sotatercept Low Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the Cmax of sotatercept in plasma.
Tmax of Sotatercept at Low Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the Tmax of sotatercept in plasma.
AUC0-inf of Sotatercept at Low Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the AUC0-inf of sotatercept in plasma.
AUC0-last of Sotatercept at Low Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the AUC0-last of sotatercept in plasma.
t1/2 of Sotatercept at Low Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the t1/2 of sotatercept in plasma.
CL/F of Sotatercept at Low Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the CL/F of sotatercept in plasma.
Vz/F of Sotatercept at Low Dose | Predose and at designated timepoints (up to approximately 120 days postdose
  Blood samples will be collected to determine the Vz/F of sotatercept in plasma.
Number of Participants who Experienced an Adverse Event (AE) | Up to approximately 120 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants who Discontinued the Study Due to an AE | Up to approximately 120 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Anaheim Clinical Trials ( Site 0007), Anaheim, California
  - Advanced Pharma CR, LLC ( Site 0005), Miami, Florida
  - QPS-MRA, LLC ( Site 0004), South Miami, Florida
  - Bio-Kinetic Clinical Applications, LLD dba QPS-MO ( Site 0003), Springfield, Missouri

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com